CLINICAL TRIAL: NCT04391244
Title: Investigating National Solutions for Personalised Iodine-131 Radiation Exposure - Measuring Absorbed Dose to Tumour and Organs at Risk Following Routine Iodine Ablation Therapy
Brief Title: Investigating National Solutions for Personalised Iodine-131 Radiation Exposure
Acronym: INSPIRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5109; 20/EM/0022 (Other: REC No)
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-04

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Radioiodine Therapy; Radiation Dose; Dosimetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-arm non-interventional prospective observational study to perform quantitative I-131 imaging and patient-specific dosimetry for patients undergoing radioiodine treatment.

DETAILED DESCRIPTION:
The hypothesis underlying this study is that treatment outcome in molecular radiotherapy is dependent on the absorbed doses delivered rather than on the radioactivity administered. For up to 50 patients, post treatment dosimetry will be performed to establish the range of absorbed doses and associated uncertainties delivered to thyroid remnants, residual disease, and healthy organs from an ablative administration of I-131 radioiodine.

Imaging systems in participating centres will be characterised (system volume sensitivity, partial-volume effect and dead-time) and set up for quantitative imaging to allow for collation of data. Patients will be assigned to one of two dosimetry gamma camera scanning schedules. For scanning schedule 1 (Standard of Care) a single standard-of-care scan (SPECT/CT) will be acquired according to local protocol with regards to time post-radioiodine administration. A minimum of 20 patients will be assigned to scanning schedule 2 (Standard of Care + Additional Imaging), for which a standard-of-care scan and two to four additional SPECT scans will be acquired between 6 - 168 hours post-administration.

SPECT imaging datasets will be reconstructed with attenuation and scatter corrections to allow quantitative dosimetry calculations. Time integrated activity will be derived from analysis of the quantitative SPECT data and combined with relevant dose factors to obtain absorbed dose estimates for each target tissue. The subset of patients with additional imaging will be used to establish the pharmacokinetic properties of radioiodine in each tissue type (biological retention half-life) to enable determination of time integrated activity in patients with a single standard-of-care scan.

A minimum of 3 whole-body retention measurements will be performed per day during the patient's stay in hospital, approximately every 2-6 hours, according to local standard of care procedures. At each external measurement time point the quantified level of radioactivity in the whole body will be recorded.

Patients will be followed-up at their standard-of-care clinic visits to assess the success of treatment as well as for short to mid-term toxicity. Results from standard of care biochemical, radiological and haematological assessments (TSH, thyroglobulin, anti-thyroglobulin antibodies, ultrasound, serum creatinine, haemoglobin, white cell count, neutrophil count and platelet count) will be recorded to assess response to treatment. Statistical analysis of the relationship between the absorbed doses and outcome data will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically proven DTC (pT1b - pT3, any N, any M)
* Total thyroidectomy performed
* WHO PS 0-2 (autonomous, self-caring)

Exclusion Criteria:

* External radiotherapy in the last 6 weeks
* Systematic chemotherapy in the last 6 weeks
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Differentiated Thyroid Cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Range of absorbed doses and associated uncertainties delivered to thyroid remnants, residual disease, metastatic disease and healthy organs. | 9 months
  To establish the range of absorbed doses and associated uncertainties delivered to thyroid remnants, residual disease, metastatic disease and healthy organs from an administration of I-131 radioiodine.

SECONDARY OUTCOMES:
Proportion of patients with successful treatment. | 9 months
  Investigation into the relationship between quantitative uptake values and/or absorbed doses delivered and treatment success. Treatment success will be defined by a thyroglobulin level of less than 2.0 ng per millilitre at 6-9 months post treatment.
Threshold absorbed dose to the thyroid remnant for treatment success. | 9 months
  To establish a threshold absorbed dose to the thyroid remnant required for treatment success. The association between these absorbed doses and the therapy outcome will be investigated, using logistic regression modelling as appropriate, with absorbed dose as a continuous variable. The relationship between the absorbed doses delivered and treatment success will be analysed using ROC analysis to establish a threshold absorbed dose for treatment success.
Association of biomarkers with absorbed dose | 9 months
  The association between absorbed doses and biomarkers (routine clinical haematological and biochemistry measurements) will be investigated using univariate logistic regression modelling as appropriate, with haematological and biochemistry measurements as continuous variables.
Association of biomarkers with treatment success | 9 months
  The association between treatment success and biomarkers (routine clinical haematological and biochemistry measurements) will be investigated using univariate logistic regression modelling as appropriate with haematological and biochemistry measurements as continuous variables. Treatment success will be defined by a thyroglobulin level of less than 2.0 ng per millilitre at 6-9 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Newbold, Study Chair — Consultant Clinical Oncologist; Glenn Flux, Principal Investigator — Head of Radioisotope Physics
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taprogge J, Abreu C, Vavrova L, Carnegie-Peake L, Rushforth D, Gape P, Gear J, Murray I, Wong KH, Newbold K, Yusuf S, Flux G. Initial results of the INSPIRE clinical trial-investigating radiation dosimetry for differentiated thyroid cancer patients. Front Nucl Med. 2023 May 15;3:964478. doi: 10.3389/fnume.2023.964478. eCollection 2023. PMID 39380954